CLINICAL TRIAL: NCT02629328
Title: CardioCel Tri-leaflet Repair Study; a Prospective, Non-randomised, Single Arm, Multi-centre Clinical Investigation
Brief Title: CardioCel Tri-leaflet Repair Study
Acronym: CTRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anteris Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRS-2015-01; EUDAMED (Other: CIV-15-07-013706)
Record Dates: First submitted 2015-11-16; First posted 2015-12-14 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Aortic Stenosis; Aortic Insufficiency
Keywords: CardioCel; FDA cleared; Tri-leaflet repair; Aortic valves
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CardioCel (Other): Treatment with CardioCel implant
  Interventions: Device: CardioCel

INTERVENTIONS:
Device: CardioCel — Treatment with CardioCel implant

SUMMARY:
This study will quantify the safety and efficacy of the CardioCel implant in tri-leaflet repair. 80 patients in up to 7 sites in Europe and the US will all be treated with the CardioCel implant.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the CardioCel for the repair of aortic valve stenosis and/or insufficiency. CardioCel is a cardiovascular patch manufactured with the so called ADAPT® technology. The ADAPT technology uses bovine spongiform encephalopathy-free pericardium which is processed in several ways to make it biocompatible with human tissue. CardioCel should provide an off the shelf material solution for tri-leaflet repair surgery due to its functional attributes, low propensity for post implant calcification, and overall biocompatibility. As a result adverse events and complications associated with the autologous pericardium repair surgery are mitigated.

In this study patients suffering from moderate-to-severe aortic stenosis and/or aortic insufficiency will be included.

In this study 80 patients will be enrolled in up to 7 centers in Europe and the US. The expected study duration is 36 months; 12 months of recruitment and 24 months follow-up.

CardioCel is US FDA cleared for the repair of cardiac and vascular defects, including intra-cardiac defects; septal defects, valve and annulus repair, great vessel reconstruction, peripheral vascular reconstruction, suture line buttressing and pericardial closure.

ELIGIBILITY:
Inclusion Criteria:

1. The subject's annular measurements are ≥ 19 mm to < 27mm as confirmed on pre-op echo and inter commissure distance equal to or bigger than 19mm as confirmed intraoperatively.
2. The subject is suitable for a tri-leaflet repair.
3. The subject has documented moderate-to-severe AS and/or AI.
4. The subject is willing and able to comply with specified follow-up evaluations, including trans oesophageal echocardiography (TEE) if there are inadequate images by transthoracic echocardiography (TTE) to assess the aortic valve. The subject has reviewed and signed the written informed consent form.
5. The subject upon final intraoperative assessment has intracardiac anatomy suitable for tri-leaflet repair using CardioCel.

Exclusion Criteria:

1. Greater than 85 years of age at the time of consent.
2. The subject's annular measurements < 19 mm or > 27mm.
3. All patients will be excluded who require emergent surgery (within 24 hours of a presentation to an emergency department) for any reason.
4. The subject will be excluded with pre-existing valve prosthesis in the aortic position.
5. Patients requiring repair of other cardiac valves will be excluded.
6. The subject has active endocarditis.
7. Heavily calcified aortic roots or "porcelain aortas" (as evidenced on cardiac echo).
8. Leukopenia with a WBC of less than 3000 cells per microliter.
9. Acute anaemia with a haemoglobin less than 8 g/dL.
10. Platelet count less than 150.000 platelets/microliter.
11. History of a defined bleeding diathesis or coagulopathy or the subject refuses blood transfusions.
12. Active infection requiring antibiotic therapy (if temporary illness, subjects may enrol 2-4 weeks after discontinuation of antibiotics).
13. Subjects in whom trans oesophageal echocardiography (TEE) is contraindicated.
14. Low Ejection Fraction (EF) < 35%.
15. Life expectancy < 1 year, or severe comorbidities, such as cancer, dialysis, or severe COPD at the investigator's discretion
16. The subject is an illicit drug user, alcohol abuser, prisoner, institutionalised, or is unable to give informed consent.
17. The subject is pregnant or lactating (non-pregnancy to be confirmed by pregnancy test for all child bearing potential females prior to enrolment).
18. Recent (within 6 months) cerebrovascular accident (CVA) or a transient ischemic attack (TIA).
19. Myocardial Infarction (MI) within one month of trial inclusion
20. Upon intraoperative assessment of the intracardiac anatomy the patient is not suitable for tri-leaflet repair using CardioCel.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-09; Primary Completion 2017-07-05 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
In-hospital survival (defined as percentage of patients alive and discharged from the index operation - presented as the inverse, or standard surgical operative mortality) | Pre-operative to 14 days post-operative
Changes in mean aortic valve gradients from preoperative (baseline screening) to 6 months post-valve repair assessed by transthoracic or transesophageal echocardiography | Pre-operative to 6 months post-valve repair
Mean transaortic valve gradient, measured using echocardiography, postoperatively, and at 6 and 12 months after valve repair. | Up to 12 months post-valve repair
Aortic regurgitation grade (assessed on a 0-4 scale), measured using echocardiography, postoperatively, and at 6 and 12 months after valve repair. | Up to 12 months post-valve repair

SECONDARY OUTCOMES:
Changes from preoperative to 6-months postoperative in linear left ventricular (LV) diastolic and systolic dimensions measured from parasternal long axis views by echocardiography. | Pre-operative to 6 months post-valve repair
Changes from preoperative to 6-months postoperative in left ventricular volume measured by the Simpson's Biplane method using echocardiography. | Pre-operative to 6 months post-valve repair
Changes from preoperative to 6-months postoperative in LV mass (if calculated), using the area-length method, assessed by echocardiography. | Pre-operative to 6 months post-valve repair
Changes in symptomatic status (NYHA CHF Classification) from preoperative to 6 months after aortic valve repair. | Pre-operative to 6 months post-valve repair
Changes in patient reported outcomes (EQ-5D) from baseline to 26 week postoperative | Baseline to 26 weeks post-valve repair
Implant procedure success (evaluated through post-procedure hospital discharge) measured by the incidence of pre-defined adverse events: | From study enrolment to 24 months post-valve repair

CONTACTS AND LOCATIONS:
Overall Officials: Dominico Mazzitelli, M.D., Principal Investigator — German Heart Centre of the Technical University
Locations (1):
- Universtiy Hospital Leuven, Leuven, Belgium